CLINICAL TRIAL: NCT02179489
Title: Randomized Multicentric Phase III Trial Comparing Simple Surgery to Surgery Plus HIPEC (Hyperthermic Intraperitoneal Chemotherapy) With MMC in Colorectal Patients Who Have a High Risk of Developing Colorectal Peritoneal Carcinomatosis
Brief Title: Surgery With HIPEC in Treating Patients With a High Risk of Developing Colorectal Peritoneal Carcinomatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Prof., Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRCCZ-C01
Record Dates: First submitted 2014-06-21; First posted 2014-07-01 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Malignant Neoplasm of Large Intestine TNM Staging Primary Tumor (T) T4; Peritoneal Carcinomatosis
Keywords: Peritoneal carcinomatosis; HIPEC; controlled clinical trial; colorectal cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Colorectal Neoplasms | interventions — Surgical Procedures, Operative; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): surgery alone
- Hipec (Experimental): Surgery and Hyperthermic Intraperitoneal Chemotherapy with MMC
  Interventions: Procedure: Surgery and Hyperthermic Intraperitoneal Chemotherapy with MMC

INTERVENTIONS:
Procedure: Surgery and Hyperthermic Intraperitoneal Chemotherapy with MMC — HIPEC with MMC: Mitomycin C (MMC) (30 mg/m2 of body surface area). Closed technique, as preferred. Duration: 60 minutes. Mean Intra-abdominal Temperature: 43°C.
  Arms: Hipec

SUMMARY:
Multicentric randomised trial. The goal of this clinical research study is to learn if hyperthermic intraperitoneal chemotherapy (HIPEC) will help to decrease the rate of peritoneal carcinomatosis(PC) in patients with high risk of developing PC of colorectal cancer. The safety of this treatment will also be studied.

DETAILED DESCRIPTION:
Hyperthermic intraperitoneal chemotherapy(HIPEC) is a recently validated option for the treatment of peritoneal carcinomatosis from colorectal or ovarian origin. This therapeutic program demonstrated a significant improvement of overall survival of the disease. It is not yet known whether surgery followed by HIPEC is effective on decreasing the rate of peritoneal carcinomatosis(PC) in patients with high risk of developing PC of colorectal cancer.Patients with a high risk of developing colorectal Peritoneal Carcinomatosis (PC), defined by Colorectal Cancer With a Resected Minimal Synchronous PC or Ovarian Metastases, or identified T4 by intraoperative pathological diagnosis, or Tumour Rupture in the Abdominal Cavity. If patients with a high risk of developing PC identified by preoperative examination, they will be informed and will sign the consent. After complete resection of their tumor, they will be randomised to surveillance alone (control group) or HIPEC (experimental group). All patients will receive the current standard postoperative adjuvant treatment : 6 months of systemic chemotherapy (currently including FOLFOX4, mFOLFOX6, CapeOx or Capecitabine regimen which could be modified if the standard is modified). Then a work-up is done to find recurrence. If the recurrence occurs, the patient will be treated with the best known treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with the following history:

  1. Histologically-proven colorectal adenocarcinoma
  2. Presenting at the time of resection of the primary with one of the following 5 criteria (criteria indicating a high risk of developing PC) :

     * Minimal PC, resected at the same time as the primary
     * Rupture of the primary tumour inside the peritoneal cavity,
     * Intraoperative rupture of the primary tumour during surgery
     * Histologically-proven T4 colorectal adenocarcinoma
* Who have received standard systemic adjuvant chemotherapy (6 months of systemic chemotherapy) :

  1. Chemotherapy with FOLFOX4, mFOLFOX6, CapeOx or Capecitabine(the current standard treatment; it can be modified in the future in the two groups, if the standard is modified)
  2. Given on an intent-to-treat basis (it can be stopped prematurely for miscellaneous reasons)
* Patients who do not present any sign of tumour recurrence at the end of these 6 months of chemotherapy
* Patients with the following general characteristics:

  1. Age between 18 and 75 years
  2. Performance Status (ECOG) 0, 1 or 2, life expectancy > 12 weeks
  3. Adequate renal, and bone marrow function: a. Leukocytes >/= 3,000/microL; b. Absolute neutrophil count >/= 1,500/microL; c. Platelets >/= 100,000/Ul; d. Serum creatinine </= 1.5 mg/dL
  4. Hepatic function: a. AST (SGOT)/ALT (SGPT) </= 5 X institutional (Upper Limit of Normal) ULN
  5. Operable patients
  6. Completion of neoadjuvant systemic chemotherapy
* Patients will be informed and a signed consent before initiating any procedure specific to the trial

Exclusion Criteria:

1. Cancers of non colorectal origin
2. Patients presenting with a detectable recurrent tumour
3. History of cancer (excepted cutaneous basal cell carcinoma or in situ carcinoma of the uterine cervix) with a recurrence during the 5 previous years
4. Known HIV, Hepatitis B or Hepatitis C positive
5. Pregnant women or likely to be pregnant
6. Persons under guardianship
7. Subjects deemed unable to comply with study and/or follow-up procedures.
8. Subjects with a known hypersensitivity to protocol systemic chemotherapy that was life-threatening, required hospitalization or prolongation of existing hospitalization, or resulted in persistent or significant disability or incapacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Three years from the date of randomization
  DFS

SECONDARY OUTCOMES:
3 year overall survival | 3 years
  3-OS
Peritoneal disease-free survival | 3 years
  PDFS
5 year overall survival | 5 years
  5-OS
morbidity | Baseline before any treatment,3 months post operation, 1 year post operation
  Toxicity induced by HIPEC using the NCI CTC criteria; one month and six months morbidity.
  Subgroup analysis: pT4; pts. ≤ 40yrs.
QOL | Baseline before any treatment,3 months post operation, 1 year post operation
  Duration of operation; return of bowel function; length of hospital stay; return to normal activity; six months and one year QOL, using the SF-36 v1.0; percentage of patients in both arms completing the scheduled postoperative chemotherapy; Subgroup analysis: pT4; pts. ≤ 40yrs.

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, Prof., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (9):
- China (9):
  - Union Hospital Fujian Medical University, Fuzhou, Fujian
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Second Affiliated Hospitalof Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - People's Hospital of Shaoxing, Shaoxing, Zhejiang
  - Yuyao People's Hospital, Yuyao, Zhejiang

IPD SHARING:
Plan to Share IPD: No